CLINICAL TRIAL: NCT05134324
Title: The Effects of rTMS and tDCS Copuled With Robotic Therapy on Upper Extremity Functional Recovery in Patients With Chronic Stroke
Brief Title: The Effects of rTMS and tDCS Copuled With Robotic Therapy In Patients With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associate professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22
Record Dates: First submitted 2021-11-11; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Chronic Stroke
Keywords: stroke; rTMS; tDCS; robotic therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- active rTMS (Experimental): Participants recevied 1 Hz low frequency repetetive TMS during 20 minutes and a total of 1200 stimuli for 15 sessions. The patient received robotic therapy for upper extremity just after each active TMS sessions
  Interventions: Other: active rTMS
- sham rTMS (Sham Comparator): Participants recevied sham TMS during 20 minutes and a total of 1200 sham stimuli for 15 sessions with sham coil. The patient received robotic therapy for upper extremity just after each sham TMS sessions
  Interventions: Other: sham rTMS
- active tDCS (Experimental): Participants recevied 2 mA anodal transcranial direct current stimulation 20 minutes for 15 sessions. The patient received robotic therapy for upper extremity just after each active tDCS sessions
  Interventions: Other: active tDCS
- sham tDCS (Sham Comparator): Participants recevied sham stimulation. The patient received robotic therapy for upper extremity just after each sham tDCS sessions
  Interventions: Other: sham tDCS

INTERVENTIONS:
Other: active rTMS — Participants recevied 1 Hz low frequency repetetive TMS during 20 minutes and a total of 1200 stimuli for 15 sessions. Motor threshold was defined as the minimum stimulus intensity eliciting 5 responses of about 50 µV out of 10 consecutive trials (50% successful MEPS) in the relaxed contralateral abductor pollicis brevis (APB).The patient received robotic therapy for upper extremity just after each active TMS sessions.
  Arms: active rTMS
Other: sham rTMS — Participants recevied sham TMS during 20 minutes and a total of 1200 sham stimuli for 15 sessions with sham coil employed was identical in shape and size to the real stimulation coil and produced no magnetic field. The patient received robotic therapy for upper extremity just after each sham TMS sessions.
  Arms: sham rTMS
Other: active tDCS — Participants recevied 2 mA anodal transcranial direct current stimulation 20 minutes for 15 sessions.The electrodes will be placed anodal to the C3/C4 (International 10/20 Electroencephalogram System) area, corresponding to the location of the affected hemisphere primary motor cortex (M1), and cathodal to the contralateral supraorbital region. The patient received robotic therapy for upper extremity just after each active tDCS sessions.
  Arms: active tDCS
Other: sham tDCS — Participants recevied sham stimulation were applied current was ramped up either over 10 seconds, with an equal amount of time for tapering off. The patient received robotic therapy for upper extremity just after each sham tDCS sessions
  Arms: sham tDCS

SUMMARY:
The purpose of this study is to assess the effect of rTMS and tDCS coupled with robotic therapy on upper extremity functional recovery

DETAILED DESCRIPTION:
After being informed about study and potential risks, all patient giving written informed consent will undergo screening period determine eligibility for study entry. The patients who meet the eligibility requirements will be randomized into four groups in a 1:1 ratio to active rTMS, sham rTMS, active tDCS and sham tDCS.

ELIGIBILITY:
Inclusion Criteria:

* ischemic stroke with a disease interval of 6 months to 2 years
* aged based 18 years
* first stroke
* Mini mental test score ≥ 22
* upper extremity (elbow, wrist and finger) spasticity level Modified Ashworth Scale (MAS)≤2
* Shoulder, elbow and wrist muscle strength ≥ 2 according to Medical Research Council- MRC

Exclusion Criteria:

* hemorrhagic stroke
* history of epilepsy
* a cardiac pacemaker
* pregnancy
* Fugl Meyer upper extremity assessment score ≥44
* history of previous stroke or ischemic attack
* neurological diseases other than stroke
* metallic implant in brain or scalp (including cochlear implant)
* previous brain surgery
* orthopedic disease that prevents upper extremity movements
* diagnosis of malignancy
* receiving robotic /TMS/tDCS treatments in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-02-25 (Estimated); Study Completion 2022-05-25 (Estimated)

PRIMARY OUTCOMES:
Upper Extremity Fugl-Meyer Motor Function Scale | initial, 3th week 9th week changes
  Scale measures level of upper extremity motor functions (min-max: 18-126 points). Higher values represent a better outcome.

SECONDARY OUTCOMES:
Motor Activity Log-28 | initial, 3th week 9th week changes
  Scale measures frequency of use and functionality level of the affected upper limb during daily activities (min-max: 0-5 points). Higher values represent a better outcome.
Barthel Index | initial, 3th week 9th week changes
  Scale measures performance in activities of daily living. The Index yields a total score out of 100 - the higher the score, the greater the degree of functional independence.
Stroke Impact Scale version 3.0 | initial, 3th week 9th week changes
  Scale has 8 domains: strength, hand function, mobility, physical and instrumental activities of daily living, memory and thinking, communication, emotion, and social participation. Scores for each domain range from 0 to 100, and higher scores indicate a better Scores for each domain range from 0 to 100, and higher scores indicate a better. The scale also includes a question (item 50) to assess the patient's global perception of recovery. The respondent is asked to rate his or her percentage of recovery on a visual analog scale of 0 to 100, with 0 meaning no recovery and 100 meaning full recovery.
Box and Block Test | initial, 3th week 9th week changes
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. Higher values represent a better outcome.
Modified Ashworth Scale | initial, 3th week 9th week changes
  Scale measures muscle tone (spasticity) (min-max:0-4). Higher values represent a worse outcome
The amplitude of motor evoked potentials (MEPs) | initial, 3th week 9th week changes
  The amplitude of MEP is a common yet highly variable measure of corticospinal excitability.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Celik Karbancioglu, MD, Study Director — SBU,Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No